# Operations Manual/Study Protocol

## STOP: Stop Smoking Therapy for Ontario Patients

# **Operations Manual and Protocol for Study Personnel**

# **Study Sponsor** Ministry of Health and Long-term Care **Pfizer Consumer Health Care**

**Centre for Addiction and Mental Health** 33 Russell Street Toronto, ON M5S 2S1

**Principal Investigator** 

Peter Selby, MBBS

(416) 535-8501 ext 6859 (office)

(416) 260.4170 (fax)

peter selby@camh.net

**Project Coordinator** 

Rosa Dragonetti, MSc

(416) 535-8501 ext 6343 (office)

(416) 260.4170 (fax)

rosa dragonetti@camh.net

Research Analyst Virginia Ittig-Deland

(416) 535-8501 ext 6762 (office)

(416) 260.4170 (fax)

virgina ittig-delan@camh.net

**Scientist** 

Laurie, Zawertailo, Ph.D.

(416) 535-8501 ext 6007(office)

(416) 595-6618 (fax)

laurie zawertailo@camh.net

**Research Assistant** 

Janet Ho, B.A.

(416) 535-8501 ext 6702(office)

(416) 260.4170 (fax)

janet ho@camh.net

**Project Secretary** 

Janey Haggart

(416) 535-8501 ext 4455 (office)

(416) 260.4170 (fax)

janey\_haggard@camh.net

Y:\Peter Selby Projects\STOP\Nonactive STOP Arms\STOP 1 CAMH MODELS\Study Operations Manual\STOP Operations Manual V9 24Mar2006.doc

# **Table of Contents**

| Study Preamble | |
|---|---|
| Study Site Information | |
| Description of NRT | 4 |
| Ordering, Tracking, packaging, preparation, dispensing Ordering Tracking Dispensing | 2<br>5 |
| Storage | 6 |
| Recruitment Recruitment. Initial Eligibility. Screening. Inclusion/exclusion Criteria. Screening/enrollment. | |
| Data Collection and Enrollment Consent Procedure. Enrollment. Initial Assessment. Lab Tests. Specimen Packaging Guidelines. Carbon Monoxide. Follow up appointments. Self-selection. | 10<br>10<br>11 |
| Treatment Protocol Deviations and Violations | 1 |
| Study Duration | 12 |
| Confidentiality | 12 |
| Dealing with Impaired Participants | 12<br>13 |
| · | |
| Dealing with Impaired Participants | 13 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. | 13<br>13 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. Non-pharmacological Treatment. | 13<br>13<br>13 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. Non-pharmacological Treatment. Training for Research Staff. | 13<br>13<br>13 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. Non-pharmacological Treatment. Training for Research Staff. Adverse Event Recording. | 13<br>13<br>13<br>13 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. Non-pharmacological Treatment. Training for Research Staff. Adverse Event Recording. Reporting Occurrences/Incidents. | 13<br>13<br>13<br>13<br>14 |
| Dealing with Impaired Participants. Hospitalization/Incarceration. Non-pharmacological Treatment. Training for Research Staff. Adverse Event Recording. Reporting Occurrences/Incidents. List of Study Forms and Attachments. Individual Study Models Protocols NRT-only Model. Treatment-as-Usual Model. Counsellor Model. Pharmacy Model. Physician Model. | 13<br>13<br>13<br>14<br>18<br>17<br>18<br>20<br>22<br>22 |

### **Study Preamble**

The purpose of this STOP Study Operations is to provide each model with the information necessary for the uniform implementation of the clinical intervention and the standardized collection of outcome data, and, in so doing, ensure consistency in keeping with ethical standards of research.

The CAMH models for STOP discussed in this manual include:

- o Treatment-as-Usual Model
- o Pharmacy Model
- o NRT-only Model
- o Physician Model
- o Nurse Model to be determined
- o Counsellor Model

### **Study sites information**

### **Centre for Addiction and Mental Health**

The STOP Study includes several sites across the province. This Operations Manual is specific to the models to be run out of the Nicotine Dependence Clinic (NDC) at CAMH. Participants recruited to the study will be seen at the NDC- Russell Street Site.

### **Description of NRT**

The nicotine replacement therapies that are used in this study include the Nicoderm patch (21, 14 and 7mg doses), the Nicorette gum (2 and 4mg) and the Nicorette inhaler. See package insert for a complete description of the products (Attachment 5).

### Ordering, tracking, packaging, preparation, dispensing

### **Ordering Initial shipments**

NRT will be ordered through the contact at Pfizer: Bill Carroll (905-968-2510) The RA and Pharmacist (Eva) will order a supply of NRT on a monthly basis from Pfizer warehouse using the NRT Order Form-Pfizer (*Appendix R*). The NRT will be stored in the pharmacy storage in the basement.

### Ordering additional NRT

The Research Assistant will track NRT stock for all treatment models and will plan to reorder additional supply of NRT 4 weeks prior to depletion of stock. The Research Assistant will consult with Pharmacy staff (Eva) before ordering next shipment to ensure that space is available for next shipment. The RA will use an NRT Order Form-Pfizer (Appendix R) to order additional supply of medication.

#### Treatment-as-Usual Model

Ss will get their NRT from the ARF Pharmacy as per usual practice. Pharmacy will use STOP NRT only for Ss subjects. During Wednesday evening clinic, the NDC nurse will dispense the NRT. The RA and NDC nurse will meet weekly to order additional NRT using the NRT Internal Order Form (Appendix S). The subjects in this model will be provided with only 10-weeks of one form of NRT from the STOP Study. Any additional NRT that a subject may use is to be prescribed or purchased outside of the realm of the study and be recorded as a concomitant medication on the Concomitant Medications Record (Appendix U).

### **NRT-only Model**

The RA will order a supply of NRT on a weekly basis from Pharmacy using the NRT Internal Order Form (Appendix S). The NRT will be stored in a locked cabinet in the RA's office. Only the RA and Scientist will have access to this cabinet.

### **Pharmacy Model**

The Pharmacy will use STOP NRT stock for Ss. Pharmacy will track the amount of NRT dispensed using their internal database.

### **Counsellor and Physician Models**

The RA will order a supply of NRT on a weekly basis from Pharmacy using the NRT Internal Order Form (Appendix S)

### Tracking: Keeping inventory/dispensation records of NRT

A **Drug Shipment Record** (*Appendix T*) will document:

- 1. Medication (indicate patch, gum, or inhaler)
- 2. Date received
- 3. Expiry date and lot number
- 4. Strength
- 5. Quantity

A **Drug Administration/Subject Record Log** (*Appendix M*) will be used to track the NRT dispensed to Ss. The log will identify:

- 1. Subject ID
- 2. Study#
- 3. Date dispensed
- 4 Dose
- 5. Type of NRT: include lot number
- 6. Dispensed by

A Concomitant Medications Record (Appendix U) will be created for each participant. The record will be stored in each subject's chart and will identify:

- 1. Medication (patch, gum, inhaler) This section is meant for drugs other than actual study drug and should capture all medications taken by the subject at the onset and duration of the study.
- 2. Dose
- 3. Frequency
- 4. Indication
- 5. Start date
- 6. Stop date

### **Dispensing the NRT**

Dispensation of the NRT for the study shall be in accordance with the **CAMH Delegation of Dispensing Policy** (*Attachment 4*).

Ss will receive a total of 10 weeks of NRT. Research staff will dispense type and dose of NRT based on approved use of the medication and will not provide off-label use. If subjects want to use a combination of NRT or increase their dose or NRT, they may do so by purchasing additional NRT at their local pharmacy. This data/information should be collected and recorded in each Ss chart. Additional use of NRT will be recorded as a Protocol Violation (see page 11).

### **Dispensing by Research Assistant**

The RA will be trained in dispensing NRT by CAMH Pharmacy staff and will store and dispense for several models of the study including the NRT-only model, the Physician Model and the Counsellor Model. The RA will also serve as back-up for other models when usual staff are unavailable. The RA will complete a **Medication Used in Research Studies Dispensation**Form (available from Pharmacy). This form will be kept in the Pharmacy with a copy in the Research Binder. The RA will maintain records of each dose dispensed using the **Drug**Administration Subject Record (Appendix M). NRT used by the RA will be kept in a locked cabinet in a locked room.

For the NRT-only Model: The RA will take Ss into a designated office, which will display the NRT on shelves. Ss will take their recommended NRT and the RA will stamp their NRT Card.

### **Dispensing by Pharmacy**

Pharmacy will maintain control records of dispensing of the research NRT. Pharmacy will use the **Drug Administration Subject Record** (*Appendix M*) to track the dispensed NRT. Pharmacy will dispense to the following models:

- Pharmacy Model
- NDC Treatment as Usual Model: Physicians will prepare the prescription using the STOP Prescription Form (Appendix Q) for the NRT and Ss will take the prescription to the Pharmacy. Pharmacy will dispense as per usual practice for CAMH clients. However, Pharmacy will track the NRT dispensed using the above forms.

### **Dispensing by Nurse**

The RNs will track the NRT dispensed using the **Drug Administration Subject Record** (*Appendix M*). Nurses will dispense the NRT for the following models:

- **Nurse Model:** The Study Nurse will dispense the NRT according to the **NRT Algorithm** (*Appendix N*).
- **NDC Treatment as Usual Model**: The NDC Nurse will dispense NRT for the clinic on Wednesday evening (4:00 7:00 p.m.).

Any additional NRT prescribed by the NDC physician will be paid for by the subject/client and will not be provided from STOP NRT stock. Any NRT that is given to Ss in addition to their 10-weeks should be recorded as protocol violations (See Section on Protocol Violation page 11).

### **Storage**

The NRT shipped to CAMH will be stored in Pharmacy's Storage area (in the basement of the East wing of 33 Russell Street site). Pharmacy will track the NRT supply and the RA will have a copy of the tracking forms. The RA will complete an internal **NRT Internal Order Form** (Appendix S) to stock local supplies (i.e., supply for different models in NDC). Local supplies of NRT will be kept in a locked cabinet in a locked room in the Nicotine Dependence Clinic. A limited number of individuals will be have access to this cabinet and these individuals will be specified in writing on the **Signature and Delegation of Authority Log** (Appendix V).

### **Returned/Unused NRT**

Some study subjects may choose to return their unused, unopened packages of NRT. This may happen if the subject has quit and no longer feels the need to use NRT. Subjects should be informed that they may want to taper off slowly before stopping the NRT completely to assess whether they may experience withdrawal once again.

If subjects do not wish to continue their NRT, you may accept their unused packages. These packages should be returned to the CAMH pharmacy to be disposed of according to appropriate procedures. Staff should document the amount, type, dose and lot number of the NRT that is being returned before giving it to the pharmacy.

Subjects may also keep their unused NRT and should be advised to consult with their physician or pharmacist if they wish to restart the NRT at a later date.

DO NOT reuse the returned the NRT for other study subjects.

### Recruitment, Enrollment

#### Recruitment

Study Subjects (Ss) will be recruited through various methods. CAMH programs will refer their clients who are interested in quitting smoking to the study. Advertisements and posters will be distributed internally at CAMH to make CAMH internal programs and staff aware of the study.

Advertisements will also be placed in local media to recruit Ss. Additional recruitment strategies will be employed based on recruitment rates. All recruitment methods will be pre-approved by REB.

**Initial Eligibility Determination:** All participants entering treatment at this site or who respond to advertisements will call the research staff for an initial telephone screening. A **Telephone Screening Form** (*Appendix A*) will be used to assess eligibility.

**Those potential participants <u>failing</u> initial screening**: All screening forms of participants failing initial screening will be kept in the back section of the "Screening Binder" and filed by alphabetical order of last name. Each time a participant agrees to be screened for the study, this binder must be checked to ensure he/she has not been previously screened. A new screening form can be completed and the old screening form should then indicate that he/she was rescreened and the outcome of the re-screening.

**Those meeting initial screening**: If a potential subject indicates interest in participating in the study and meets the initial screening, a copy of the screening form is placed in front section of the "Screening Binder". Research staff will use the **Triage Form** (Appendix B) to help subjects choose the study model. The research staff will then set up an appointment with the Research Assistant (approximately 70 minutes) for the participant to sign the **Consent Form** (Appendix C) and complete the **Initial Study Assessment** (Appendix D). Other appointments (depending on study model) will be set up at this time as well.

If a potential participant is not currently in treatment and fails initial eligibility or is no longer interested in the study, he/she will be provided with a list of providers to contact for possible treatment as well as other resources that are available for smoking cessation.

### Screening

Research staff will screen potential participants using the following criteria:

### **Inclusion Criteria**

- □ Age: 18 years or older
- Ontario residents
- Current daily smoker
- $\square$  Smokes  $\ge 10$  cigarettes/day
- □ Smoked more than 100 cigarettes in their lifetime
- □ Wants to quit within next 30 days

### **Exclusion Criteria**

- □ Have a medical condition that would make participation medically hazardous as determined by the Study Physician (e.g., recent cardiovascular incident)
- □ Intolerant to NRT
- □ Have an acute severe psychiatric condition in need of immediate treatment or be an imminent risk to self or others. These subjects will be referred to a hospital emergency or the ER at the Clarke Site.

### **Subject Screening/Enrollment Log**

Research staff will track screening on the **Subject Screening/Enrollment Log** (*Appendix E*). The items to be recorded include subject initials, screen date, meets criteria (yes/no), date of enrollment into study, date declined and rationale. This form is to be kept in the Research Binder.

### **Data Collection Procedures**

#### **Consent Procedures:**

**Consent forms** (*Appendix C*) will be filed in the Research Binder. All versions will be kept in the binder and the most recent version will be filed in front of other versions. All versions of consent forms will also be stored on the T-drive. A **Consent Versions Tracking form** (*Appendix F*) found in the Research Binder will also track versions of the consent form.

- a) The research staff will escort the participant to a private office and begin the consent process.
- b) All participants will first be given a copy of the consent form and asked to follow along on her copy as the consent form is read to him/her. Prior to reading, research staff will give a general overview of the study. The potential participant will also be encouraged to ask questions about any part she does not understand as the consent form is read to her.
- c) In order to further facilitate questions, at the end of each page, and in natural breaks in the consent form section, research staff will ask if the participant has any questions. The participant will also be reminded that he/she may ask questions at any time during the consent process.

- d) Following reading of the consent form, the research staff member will ask the participant if he/she wants to participate in the study. If she does, the participant and research staff member will sign and date all copies of the consent.
- e) The research staff and the study subject will initial each page of the consent form to document review of that page.
- f) Person obtaining consent will document process and outcome, noting time of signature in the source documents.
- g) The subject will be given a copy of the signed consent form to take home.
- h) Genetics Sub-study: If Ss wish to participate in the genetics sub-study, they will provide their consent by checking off this box in the Agreement to Participate section of the study consent from and initialing it. If they consent to this sub-study, they will be administered additional questionnaires and DNA information will be collected from their blood sample.

#### **Enrollment**

After consent has been obtained, the research staff will assign a **Participant Study Code** to the initial assessment form. Research Staff will maintain a master list of the Participant Study Codes and the names of clients in the **Master Subject Study Codes** (*Appendix G*). This master list will be stored on a non-networked computer and password protected.

### **Initial Assessment Appointment**

The research staff will administer the **Initial Study Assessment** (*Appendix D*) Participants will not self-administer the questionnaires. The approximate time needed to complete the form is 45 minutes.

### Determining eligibility according to major health concerns

The Study Physician will review the medical information on each assessment on a weekly basis to determine if subjects that have special medical issues or concerns should be excluded from participating in the study.

### **Genetics Study**

For Ss that consented to participate in the genetics component of the study, they will also be administered the M.I.N.I. (Mini-International Neuropsychiatric Interview – *Attachment 1*). This will take an additional 15 to 20 minutes.

### Lab tests

Upon completion of the consent process and the Initial Study Assessment, research staff will collect blood samples from the Ss. A second sample of blood will be taken at Week 6 of the study. These biological samples will be used to determine plasma concentrations of nicotine and the main metabolites cotinine and 3-hydroxycotinine.

### **Blood:**

Purpose:

- 1. For genotyping if study subject consents
- 2. For initial plasma cotinine

Only qualified research staff who have received a certificate in venipuncture procedures will collect a blood sample from Ss.

### **Procedure for Venipuncture and Blood Handling:**

Refer to the LN.E.1 Venipuncture Procedure – (*Attachment 2*).

### **Specimen Packaging Guidelines**

To ensure patient confidentiality all specimens are to be packaged as follows:

- All containers (e.g. blood tubes) must be checked for cracks before filling and only intact containers used.
- Check that the caps and lids on all containers are secure before packaging.
- Place each specimen in a brown paper bag and close the bag.
- Requisitions are placed in the brown paper bag with the specimen(s).
- Place a label containing the proper address on the brown paper bag.

### **Tracking laboratory specimens**

All specimens collected will be tracked using the **Laboratory Specimen Tracking/Shipping Log** (*Appendix H*). The research staff will fill in the visit number, date shipped, shipping # and frozen/ambient. The **Laboratory Specimen Tracking/Shipping Log** will be kept in the Research Binder.

*Carbon Monoxide*: Research staff will use a carbon monoxide monitor to measure CO levels in participants.

The interviewer will tell the participant the following:

"I am now going to measure the level of carbon monoxide present in your body. This is going to serve as a baseline measure of your exposure to CO. CO is produced in your body in small amounts, but it is also a by-product of smoking."

### Procedure:

- 1. Research staff trained by the Laboratory or RN of the Nicotine Dependence Clinic may perform this procedure.
- 2. Turn the Smokerlyzer on using the ON/OFF switch (a short beep will be heard).
- 3. Insert the Sampling Assembly into the Sensor Housing on the Smokerlyzer.
- 4. Fit a Disposable Cardboard Mouthpiece into the clear end of the Sampling Assembly.
- 5. As long as the Smokerlyzer registers less than 5 ppm CO, press the 'Zero' button until 'GO' is displayed.
- 6. Ask the participant to inhale deeply and hold their breath. At the same time press the 'GO' button on the Smokerlyzer which will begin a 15-second count down until testing time.
- 7. Hand the Smokerlyzer to the participant.
- 8. Near the end of the 15-second count down the Smokerlyzer will beep several times ending with one long beep indicating that it is time for the participant to exhale into the cardboard mouthpiece.
- 9. When the display reads 0, have the participant exhale gently and steadily (until their lungs are emptied) into the mouthpiece making sure that a tight seal is made by the lips around the mouthpiece.
- 10. Record the date and breath CO reading (in ppm) on the initial assessment form.

- 11. Remove the Cardboard Mouthpiece from the Sampling Assembly and discard it.
- 12. To reuse press "go" again, then "zero" again and repeat the test from step 9.
- 13. Wait until the Smokerlyzer registers less than 5 ppm before performing another test.
- 14. Should problems arise during the testing process (error message "Err" or "Neg" appearing on the display) please contact the RN of the Nicotine Dependency Programs or the Laboratory for assistance.

### 6-week follow up appointment

Ss will be asked to come in to complete the 6-week Follow Up Interview (Appendix I) and to provide a blood sample. As informed consent is ongoing, determine and document that the Ss is willing to continue as a study participant. Carbon monoxide levels will also be collected.

#### **End-of-treatment assessment**

Ss will be asked to come in to complete the **End-of-treatment assessment** (Appendix J). Carbon monoxide levels will also be collected.

### Follow up assessments 3, 6, 12 months

Ss will be asked to complete a follow up assessment at 3, 6 and 12 months post-treatment. The Research staff will contact the Ss by telephone and arrange a time to complete the interview using the follow up assessments (*Appendix K*). A sub-sample of Ss will be asked to come in to provide a blood sample.

### **Self-selection**

During the initial assessment, Ss who qualify for participation in the study will be administered the **Triage Form** (*Appendix B*) to help determine which model they wish to join. The models available for subjects include:

**NRT-only Model**: Subjects receive 10 weeks of NRT approximately every two weeks and get no additional support or interventions. Refer to Page 17 for detailed procedures.

**Treatment as Usual Model**: Subjects receive 10 weeks of NRT. They are registered as CAMH clients and complete the General Assessment. They attend the Nicotine Dependence Clinic and discuss a treatment plan with their health care provider. Refer to Page 18 detailed procedures.

**Counsellor Model**: Subjects receive 10 weeks of NRT. They are scheduled to see a counselor in the Nicotine Dependence Clinic for three brief counseling sessions. Refer to Page 20 for detailed procedures.

**Pharmacist Model**: Subjects receive 10 weeks of NRT. They are scheduled to see a Pharmacist in the ARF Pharmacy for three brief counseling sessions. Refer to Page 22 for detailed procedures.

**Physician Model**: Subjects receive 10 weeks of NRT. They are scheduled to see a Physician in the Nicotine Dependence Clinic for three brief counseling sessions. Refer to Page 24 for detailed procedures.

**Nurse Model**: Subjects receive 10 weeks of NRT. They are scheduled to see a Nurse in the Nicotine Dependence Clinic for three brief counseling sessions. Refer to Page 26 for detailed procedures.

### **Treatment Protocol Deviations and Violations**

Protocol Deviations and violations are terms used interchangeably and refer to the same thing. Briefly, a protocol deviation or violation is any procedure that was not completed in the way or at the time or in the sequence that it was supposed to according to the protocol.

If a protocol violation occurs, the clinician or clinic staff will alert the RA. The RA will record the violation in the subjects chart and inform the Scientist. The Scientist will provide a weekly report to the REB and/or Research Office informing them of protocol violations. If it becomes apparent that a part of the protocol is being violated on a regular basis, then the study team will discuss possible solutions and will apply to the REB for an amendment to the protocol that will reflect these changes.

### **Study Duration**

Study participants will have access to 10 weeks of NRT. Clients will be asked to complete follow up questionnaires at 6 weeks, end-of-treatment and at 3 months, 6 months and 12 months. The follow up assessments will be conducted via the telephone. However, a sub-set of study subjects will be scheduled to come in to provide blood samples. Once participants have completed their 10-week supply of NRT, they will be advised of treatment options/programs in their community.

#### **Premature Termination or Withdrawal**

Subjects may experience adverse events due to the transdermal nicotine replacement therapy. The most serious adverse reaction associated with transdermal nicotine replacement therapy is localized itching at the site of application. If this occurs, Ss will be advised that this reaction is not serious and can be treated with aloe/lotion or cortisone-based cream as recommended by their family physicians or Study Physician. If subjects are not able to tolerate the reaction, they may voluntarily withdraw from the study at any time and for any reason. Ss may also switch to another form of NRT after consultation with the Study Scientist.

### **Missed Appointments**

Ss may miss up to three appointments. Clinicians may call the Ss after each missed appointment to reschedule. Each time the clinician calls, the Ss should be informed they will have a limited number of rebookings before they are dropped from the study. Clinicians should use the following script as a guideline when making the phone calls.

Hi (name of subject). This is (name of clinician) from the STOP study. You missed your appointment today. Are you still interested in participating in the study?

If no: Ask Ss why?? – should we do this or should Janet just follow up?

If yes: I would like to reschedule your appointment. However, I should inform you that you may not miss more than 3 appointments before you are excluded from the study. Are you available....

### **Confidentiality**

Study participants will be assigned a Participant Code and subject initials to protect confidentiality. Since a component of the study involves assessing health card utilization following study participation, the participants will provide their OHIP numbers. Research staff will maintain a confidential, password-protected database that links the participant code to the OHIP numbers

*Protecting data*: Data will be stored in computerized files that are not networked and will be password-protected. Hard copies will also be kept in locked filing cabinets in the research staff's office in the Nicotine Dependence Clinic.

*Transferring data*: A diskette and/or CD will be used to transfer the data. E-mail will be used to transfer anonymous data only where applicable and appropriate. Data transfer will occur between any of the investigators, study staff or study sites.

At the end of the study, all data will be entered into a common anonymized computerized database. All paper records will be anonymized and stored for 10 years. The Principal Investigator and delegates will have access to the data.

### **Dealing with Impaired Participants**

Study staff will refer impaired clients to the Addiction Medicine Clinic if subjects are seriously impaired. The appointment will be rescheduled.

### Hospitalization/Incarceration During Study Duration

Subjects who are incarcerated during the study will be withdrawn. Subject hospitalized during the study will be reassessed for participation. If no interruption occurs to their study protocol, they may remain in the study.

### Non-pharmacological Treatment

Ss may be referred to other treatment programs if they want additional treatment such as individual counseling or group counseling. If Ss are interested in accessing services of the Nicotine Dependence Clinic, Ss will be referred to the Assessment Department to complete a CAMH general assessment and to register as a CAMH client. Clients who want other referrals will be given a list of available resources in their community.

### **Training for Research Staff**

Research staff will attend training to use the CO Monitor, centrifuge equipment and venipuncture procedures. CO monitor training will be provided by the RN in the Nicotine Dependence Clinic. Venipuncture training will be provided by CAMH. Centrifuge training will be provided by the NDC nurse

### **Adverse Event Recording**

Y:\Peter\_Selby\_Projects\STOP\Nonactive STOP Arms\STOP 1 CAMH MODELS\Study Operations Manual\STOP Operations Manual V9 24Mar2006.doc

**Adverse Drug Reaction (ADR):** any noxious and unintended response to a drug that is caused by the administration of any dose of the drug.

**Serious Adverse Drug Reaction:** Adverse drug reaction that requires in-patient hospitalization or prolongation of existing hospitalization, that causes congenital malformation, that results in persistent or significant disability or incapacity, that is life-threatening or that results in death.

**Serious Unexpected Adverse Drug Reaction:** Serious adverse drug reaction that is not identified in nature, severity or frequency in the risk information set out in the investigator's brochure or on the label of the drug. These events are subject to expedited reporting to Health Canada under the marketed drugs AE notice.

**Adverse Event:** Adverse occurrence in the health of a clinical trial subject who is administered a drug that may or may not be caused by the administration of the drug, and includes adverse drug reaction.

Adverse Events will be reported to the Principal Investigator and Scientist immediately and will be tracked using the **Adverse Events Tracking From** (*Appendix W*) found in the Research Binder. The staff person collecting the information about the adverse event from the Ss will use the Adverse Events Form (Appendix X) which will be found in every Ss files.

### **Reporting Occurrences/Incidents**

CAMH Occurrence/Incident Reports: Research staff will complete the online Occurrence/Incident Report form for all incidents. Incident reports are filled in whenever a CAMH staff member is injured in any way or there is a near miss. These reports are required by law.

**Occurrences** are defined as: An unexpected occurrence involving the death or serious physical or psychological injury or risk thereof (near miss). Injury does not have to have occurred. The potential for injury and/or property damage (financial loss) is sufficient for an occurrence to be considered an incident.

A **Sentinel event** most often identifies a rare, adverse or potentially avoidable occurrence that has the potential to result in:

- Significant threat to patients, residents, employees, volunteers or visitors
- Imminent litigation
- Significant financial loss
- Significant damage to the reputation of the corporation.

Refer to the following link for CAMH's policy on Occurrence/Incident Reports. <a href="http://insite.camh.net/policies/policies/pc\_1\_15\_1\_occurrence\_incident\_reporting\_sentinel\_event\_pdf">http://insite.camh.net/policies/pc\_1\_15\_1\_occurrence\_incident\_reporting\_sentinel\_event\_pdf</a>

If you are unsure whether an incident or occurrence is reportable, please follow up with the Project Manager and/or Scientist. The following link will direct you to the online forms. https://home.camh.net/incidentreport/create.php

### **Study Forms**

- A. Telephone Screening Form
- B. Triage Form
- C. Consent Form
- **D.** Initial Study Assessment
- E. Subject Screening Enrollment Log
- F. Consent Versions Tracking Form
- G. Master Subject Study Codes
- H. Laboratory Specimen Tracking/Shipping Logs
- I. 6-week follow up assessment
- J. End-of-treatment Assessment
- K. 3-month, 6-month, 12-month follow up assessment
- L. Voucher Card
- M. Drug Administration Subject Record
- N. NRT Algorithm
- O. Stop Study Medication Profile
- P. STOP Progress Note
- Q. STOP Prescription
- R. NRT Order Form-Pfizer
- S. NRT Internal Order Form
- T. Drug Shipment Record
- **U.** Concomitant Medications Record
- V. Signature and Delegation of Authority Log
- W. Adverse Events Tracking Form
- X. Adverse Events Form
- Y. Suspect Adverse Reaction Report
- Z. Pharmacy Card
- AA. Quality Control Form
- **BB.** Running Balance Inventory

### **Attachments**

- 1. M.I.N.I.
- 2. LN.E.1 Venipuncture Procedure
- 3. STOP Brief Intervention Form
- 4. CAMH Delegation of Dispensing Policy
- 5. NRT Package Inserts
- 6. Cessation Resource List

# **Individual Study Models Protocols**

NRT-only Model Treatment-as-usual Model Counsellor Model Pharmacist Model Physician Model Nurse Model

### **NRT-only Model**

The NRT only model will resemble a convenience store model. Ss will be able to walk into a venue whereby NRT is displayed and Ss are permitted to choose the type and dose of NRT they wish to use. However, Ss will be instructed that they may only use one type of NRT at a time and the dose must be in compliance with package guidelines (i.e., no off-label use). No additional support will be provided in this model to emulate the experience of purchasing NRT in a convenience store. Ss are permitted to seek additional support on their own outside of the study. Such data will be recorded in the Ss file.

### Recruitment

Ss will be recruited according to STOP Operations Manual procedures. The RA will use the **Triage Form** (*Appendix B* to help subjects choose a model. Ss who are interested in receiving NRT only with no additional support may choose this model.

### **Dispensing**

Upon completion of the initial assessment, the research staff will give Ss a **Voucher Card** (*Appendix L*) to use to obtain their NRT from the study. Ss will attend the clinic bi-weekly (or as convenient), present their vouchers to the Research staff and choose the NRT for the next two weeks. Subjects may choose the type of NRT they prefer and the dose they feel is appropriate. However, they will only receive a total of 10 weeks of treatment.

Ss will be able to pick up their NRT during the following hours: Mondays 9:00 a.m. to 5:00 p.m., Tuesdays 9:00 a.m. to 5:00 p.m., Wednesdays 12:00 p.m. to 7:00 p.m., Thursdays 9:00 a.m. to 5:00 p.m. and Fridays 9:00 a.m. to 5:00 p.m.

### **Storage**

Research staff will stock NRT in a locked cabinet in a research office in the Nicotine Dependence Clinic and will keep track of the stock using the appropriate tracking forms **Drug Administration Subject Record** (*Appendix M*). The Ss will visit an office where NRT is stocked similar to a Convenience store (on shelves).

### **Termination**

The RA will schedule an appointment to complete the 10-week follow up appointment or end-of-treatment assessment. All Ss will be given a list of resources (Attachment 6) for additional support in quitting smoking. If Ss wish to attend the Nicotine Dependence Clinic at CAMH, they should be referred to general assessment to register as a CAMH client and complete a general assessment.

### **Treatment-as-Usual Model Protocol**

Subjects who wish to access the Nicotine Dependence Clinic at CAMH will be referred to this model. Subjects must register as CAMH clients and receive a Health Record Number to participate in this model.

### Recruitment

Ss will complete their general addiction assessment and nicotine assessment with the CAMH clinical staff. Nicotine Clinical staff will inform clients about the STOP study. If clients are interested, clinicians will contact the STOP research staff provide the client health record number and phone number.

Alternatively, Ss will be recruited via advertisements. Ss will call the RA to qualify for the study. The RA will use the **Triage Form** (*Appendix B*) to help subjects choose a model. Ss who wish to participate in this model will be referred to a Counsellor for a CAMH general assessment. They will also be given an appointment with an NDC Physician for a medical appointment.

### **Dispensing NRT**

### **Dispensing and Tracking**

Policy (Attachment 3). Ss will receive a total of 10 weeks of NRT. Research staff will dispense type and dose of NRT based on approved use of the medication and will not provide off-label use. If Ss are prescribed combination of NRT or dosing above approved indications, they may purchase the additional NRT. This data/information should be collected and recorded in each Ss chart. Additional use of NRT will be recorded as a Protocol Violation (see page 11). Ss may apply for an NDC subsidy if they cannot afford to pay for additional NRT prescribed by the NDC Physician. Ss may be referred to an NDC clinician to complete a subsidy form.

### **Dispensing by Pharmacy**

Pharmacy will maintain control records of dispensing of the research NRT. Pharmacy will use the **Drug Administration Subject Record** (Appendix M) to track the dispensed NRT. Physicians will prepare the prescription using the **STOP Prescription Form** (Appendix Q) for the NRT and Ss will take the prescription to the Pharmacy. Pharmacy will dispense as per usual practice for CAMH clients. However, Pharmacy will track the NRT dispensed using the above forms.

### **Concomitant Medications**

Pharmacists will use the **STOP Study Medication Profile** (*Appendix O*) form to record other medications used by the Ss during their participation in the study. This also includes any additional NRT purchased by the subject. This form is used by pharmacists as part of treatment-as-usual. Pharmacists see clients immediately following a nicotine assessment to review concomitant medications.

### **Treatment Plan**

A treament plan will be developed by the clinician for the client as per usual standard of practice of the Nicotine Dependence Clinic. The research staff will contact the client before their physician appointment to have client sign consent form and collect blood samples and complete the **Initial Assessment**. Clients will attend treatment as usual. Research staff will contact clients at 6 weeks to complete **6-week Follow Up Interview** (Appendix K) and collect a final blood sample. Clinical staff will use the **STOP Progress Note** (Appendix P) to record visits with the subjects. Ss will be seen bi-weekly. Physicians will use the **STOP Prescription Form** (Appendix Q) to prepare prescriptions for these Ss. They may prescribe combination NRT or off-label prescribing as this is the protocol used in NDC. However, STOP will only provide 10 weeks of one type of NRT. Additional NRT dispensed will be recorded in the charts and recorded as Protocol Violations (Page 11).

### Payment for medication

Ss may apply for an NDC bursary to help pay for the additional NRT they are prescribed. Ss should be referred to NDC clinicians to apply for a bursary.

### **Termination**

The RA will schedule an appointment to complete the 10-week follow up appointment or end-of-treatment assessment. Ss who require additional support may continue to attend the clinic and access treatment.

### **Counsellor Model**

The Counsellor Model will offer Ss brief interventions for smoking cessation based on the US Department of Public Health and Human Services Guidelines. The Ss will attend 3 sessions with a trained smoking cessation counselor. The counselor will follow the **STOP Brief Interventions Protocol** (*Attachment 3*).

The Study counselor will have received an orientation training to brief interventions and to the Study Protocol. In addition to procedures outlined in this section, the Counsellor will be familiar with all components of this Operations Manual. Any questions about the study procedures should be directed to the Project Scientist or the Project Manager.

Research staff will complete the initial assessment with the Ss. Ss will then be referred to the Counsellor to discuss a plan. The Counsellor will provide counseling according to the **STOP Brief Interventions Protocol** (*Attachment 3*). Ss will return at 6-weeks for a follow-up including providing blood/urine sample and CO. Subjects will come in for their initial assessment, one week post-quit date, six weeks after initial assessment and at end-of-treatment (10 weeks).

### Recruitment

Ss will be recruited according to STOP Operations Manual procedures. The RA will use the **Triage Form** to help subjects choose a model. Ss who wish to see a Counsellor for brief interventions will be referred to this model.

### **Dispensing NRT**

### **Dispensing and Tracking**

Dispensation of the NRT shall be in accordance with the CAMH Delegation of Dispensing Policy (Attachment 4). The RA will dispense the NRT and will track the NRT dispensed by completing a Drug Administration Subject Record (Appendix M). Study Subject charts will be kept in the RA's office.

### **Concomitant Medications**

The RA will collect this information at time of initial assessment and at each follow up appointment.

### **Brief Treatment Protocol**

Please see the **Brief Intervention Protocol** (*Attachment 3*) attached for complete details. Ss will be seen by the RA for an initial assessment and referred to the Counsellor if they choose the Counsellor Model. The Counsellor will see the Ss according to the schedule below:

#### Visit #1:

During this first visit, the Counsellor will help Ss determine the type and dose of NRT using the STOP NRT Algorithm (Appendix N). The Ss can change the type of NRT or dose if they choose. The Counsellor will record all changes to NRT using the Progress Note (Appendix P). During this visit, the Counsellor will also record other medications the Ss are taking using the

STOP Study Medication Profile (Appendix O). The Counsellor will use the **Brief Intervention Protocol** (Attachment 3) to collect relevant data and provide brief counseling. Ss will be asked to set a quit date during this visit and they will be given their NRT. The amount of NRT will depend on when they have set their quit date (i.e. enough NRT to last until second visit). However, the Counsellor will attempt to limit the NRT dispenses at this time to two weeks to encourage Ss to set a quit date within that time.

### **Visit #2:**

The second visit will occur within one to two weeks of their quit date. Staff can follow the treatment protocol and collect appropriate data. During this session, staff will schedule a third and final visit. Staff will also schedule approximately ½ hour with the RA. To do this, please call Janey Haggart at 4455 or Janet Ho at 6702 and ask to book a 6-week follow-up assessment.

#### **Visit #3:**

The third visit will be scheduled for 6 weeks after the Ss start NRT. Ss will be given the remaining 4 weeks of NRT. If Ss require ongoing support, they may be referred to other resources.

### **Termination**

The RA will schedule an appointment to complete the 10-week follow up appointment or end-of-treatment assessment. All Ss will be given a list of resources (*Attachment 6*) for additional support in quitting smoking. If Ss wish to attend the Nicotine Dependence Clinic at CAMH, they should be referred to general assessment to register as a CAMH client and complete a general assessment.

### **Study Forms relevant to this Model**

Brief Intervention Protocol (Attachment 3)
Cigarette Withdrawal Scale
Appointment Calendar
NRT Algorithm (Appendix N)
Pharmacy card (Appendix Z)
Drug Administration Subject Record (Appendix M)
STOP Progress Note (Appendix P)
STOP Medication Profile (Appendix O)
Adverse Events Form (Appendix N)
Smoking Cessation Resource List (Attachment 6)

### **Pharmacy Model Protocol**

The Pharmacy Model will offer Ss brief interventions for smoking cessation based on the US Department of Public Health and Human Services Guidelines. The Ss will attend 3 sessions with one of three ARF Pharmacists. The Pharmacists will follow the **STOP Brief Interventions Protocol** (*Attachment 3*).

Pharmacy staff have received an orientation training to brief interventions and to the Study Protocol. In addition to procedures outlined in this section, Pharmacists will be familiar with all components of this Operations Manual. Any questions about the study procedures should be directed to the Project Scientist or the Project Manager.

Research staff will complete the initial assessment with the Ss. Ss will then be referred to the ARF Pharmacy (make a 15-30 minute appointment with Pharmacy staff) to discuss a plan with the pharmacist. Pharmacy staff will provide counseling according to the **STOP Brief** Interventions Protocol (Attachment 3) to the Ss.

Ss will be informed they can schedule appointments with the pharmacist during the following hours:

Mondays 9:00 a.m. to 3:30 p.m.
Tuesdays 9:00 a.m. to 11:30 a.m.
Wednesdays 9:00 a.m. to 3:30 p.m.
Thursdays 9:00 a.m. to 11:30 p.m.

### Recruitment

Ss will be recruited according to STOP Operations Manual procedures. The RA will use the **Triage Form** to help subjects choose a model. Ss who wish to see a Pharmacist for brief interventions will be referred to this model.

### **Dispensing NRT**

### **Dispensing and Tracking**

Dispensation of the NRT shall be in accordance with the CAMH Delegation of Dispensing Policy (Attachment 4). The pharmacist will dispense the NRT during the hours listed above. Ss will be given a Pharmacy Card (Appendix 2) which they are to present at each visit so that the Pharmacist may record the information on the card. The information includes visit number, type and dose of NRT. Pharmacy staff will track the NRT dispensed using the database already employed by the ARF Pharmacy. They will also complete a Drug Administration Subject Record (Appendix M) Study Subject charts will be kept in the Pharmacy area in a locked folder provided by STOP and will be returned to Janet Ho when the subject completes 10 weeks.

### **Concomitant Medications**

Pharmacy staff will use the STOP Study Medication Profile (*Appendix O*) form to record other medications used by the Ss during their participation in the study. This also includes any additional NRT purchased by the subject.

### **Brief Treatment Protocol**

Please see the **Brief Intervention Protocol** (Attachment 3) attached for complete details. Ss will be seen by the RA for an initial assessment and referred to Pharmacy if they choose the Pharmacy Model. Pharmacy will see the Ss according to the schedule below:

#### Visit #1:

During this first visit, the Pharmacist will help Ss determine the type and dose of NRT using the STOP NRT Algorithm (Appendix N). The dose and type of NRT will be recorded on the Pharmacy Card. The Ss can change the type of NRT or dose if they choose. Pharmacy will record all changes to NRT using the Progress Note (Appendix P). During this visit, Pharmacists will also record other medications the Ss are taking using the STOP Study Medication Profile (Appendix O). Pharmacists will use the Brief Intervention Protocol (Attachment 3) to collect relevant data and provide brief counseling. Ss will be asked to set a quit date during this visit and they will be given their NRT. The amount of NRT will depend on when they have set their quit date (i.e. enough NRT to last until second visit). However, Pharmacists will attempt to limit the NRT dispenses at this time to two weeks to encourage Ss to set a quit date within that time.

### **Visit #2:**

The second visit will occur within one to two weeks of their quit date. Staff can follow the treatment protocol and collect appropriate data. During this session, staff will schedule a third and final visit. Staff will also schedule approximately ½ hour with the RA. To do this, please call Janey Haggart at 4455 or Janet Ho at 6702 and ask to book a 6-week follow-up assessment.

#### **Visit #3:**

The third visit will be scheduled for 6 weeks after the Ss start NRT. Ss will be given the remaining 4 weeks of NRT. If Ss require ongoing support, they may be referred to other resources.

#### **Termination**

The RA will schedule an appointment to complete the 10-week follow up appointment or end-of-treatment assessment. All Ss will be given a list of resources (*Attachment 6*) for additional support in quitting smoking. If Ss wish to attend the Nicotine Dependence Clinic at CAMH, they should be referred to general assessment to register as a CAMH client and complete a general assessment.

### **Study Forms relevant to this Model**

Brief Intervention Protocol (Attachment 3)
Cigarette Withdrawal Scale
Appointment Calendar

NRT Algorithm (Appendix N)
Pharmacy card (Appendix Z)
Drug Administration Subject Record (Appendix M)
STOP Progress Note (Appendix P)
STOP Medication Profile (Appendix O)
Adverse Events Form (Appendix N)
Smoking Cessation Resource List (Attachment 6)

### **Physician Model Protocol**

The Physician Model will offer Ss brief interventions for smoking cessation based on the US Department of Public Health and Human Services Guidelines. The Ss will attend 3 sessions with the Study Physician. The SP will follow the **STOP Brief Interventions Protocol** (*Attachment 3*).

The SP will have received an orientation training to brief interventions and to the Study Protocol. In addition to procedures outlined in this section, the SP will be familiar with all components of this Operations Manual. Any questions about the study procedures should be directed to the Project Scientist or the Project Manager.

Research staff will complete the initial assessment with the Ss. Ss will then be referred to the SP to discuss a plan. The SP will provide counseling according to the **STOP Brief Interventions Protocol** (*Attachment 3*). Ss will return at 6-weeks for a follow-up including providing blood/urine sample and CO. Subjects will come in for their initial assessment, one week post-quit date, six weeks after initial assessment and at end-of-treatment (10 weeks).

The Study Physician (SP) will see study subjects (Ss) during a designated clinic in NDC.

### Recruitment

Ss will be recruited according to STOP Operations Manual procedures. The RA will use the **Triage Form** to help subjects choose a model. Ss who wish to see a Physician for brief interventions will be referred to this model.

### **Dispensing NRT**

### **Dispensing and Tracking**

Dispensation of NRT shall be in accordance with the CAMH Delegation of Dispensing Policy (Attachment 4). The RA will dispense and track the NRT dispensed by completing a Drug Administration Subject Record (Appendix M). Study Subject charts will be kept in the RA's office.

### **Concomitant Medications**

The RA will collect this information at time of initial assessment and at each follow up appointment.

### **Brief Treatment Protocol**

Please see the **Brief Intervention Protocol** (Attachment 3) attached for complete details. Ss will be seen by the RA for an initial assessment and referred to the Physician if they choose the Physician Model. The Counsellor will see the Ss according to the schedule below:

### Visit #1:

During this first visit, the SP will help Ss determine the type and dose of NRT using the **STOP NRT Algorithm** (*Appendix N*). The Ss can change the type of NRT or dose if they choose. The SP will record all changes to NRT using the **Progress Note** (*Appendix P*). During this visit, the

Counsellor will also record other medications the Ss are taking using the STOP Study Medication Profile (Appendix O). The SP will use the **Brief Intervention Protocol** (Attachment 3) to collect relevant data and provide brief counseling. Ss will be asked to set a quit date during this visit and they will be given their NRT. The amount of NRT will depend on when they have set their quit date (i.e. enough NRT to last until second visit). However, the SP will attempt to limit the NRT dispenses at this time to two weeks to encourage Ss to set a quit date within that time.

#### **Visit #2:**

The second visit will occur within one to two weeks of their quit date. Staff can follow the treatment protocol and collect appropriate data. During this session, staff will schedule a third and final visit. Staff will also schedule approximately ½ hour with the RA. To do this, please call Janey Haggart at 4455 or Janet Ho at 6702 and ask to book a 6-week follow-up assessment.

#### **Visit #3:**

The third visit will be scheduled for 6 weeks after the Ss start NRT. Ss will be given the remaining 4 weeks of NRT. If Ss require ongoing support, they may be referred to other resources.

### **Termination**

The RA will schedule an appointment to complete the 10-week follow up appointment or end-of-treatment assessment. All Ss will be given a list of resources (Attachment 6) for additional support in quitting smoking. If Ss wish to attend the Nicotine Dependence Clinic at CAMH, they should be referred to general assessment to register as a CAMH client and complete a general assessment

### **Study Forms relevant to this Model**

Brief Intervention Protocol (Attachment 3)
Cigarette Withdrawal Scale
Appointment Calendar
NRT Algorithm (Appendix N)
Pharmacy card (Appendix Z)
Drug Administration Subject Record (Appendix M)
STOP Progress Note (Appendix P)
STOP Medication Profile (Appendix O)
Adverse Events Form (Appendix N)
Smoking Cessation Resource List (Attachment 6)

### **Nurse Model Protocol**

Currently, there is no Nurse Model. Future consideration will be given to this model.

# **Appendices**

| <b>A.</b> | Telephone Screening Form |
|-----------|-------------------------------------------------|
| <b>B.</b> | Triage Form |
| C. | Consent Form |
| D. | <b>Initial Study Assessment</b> |
| E. | Subject Screening Enrollment Log |
| F. | <b>Consent Versions Tracking Form</b> |
| G. | Master Subject Study Codes |
| Н. | Laboratory Specimen Tracking/Shipping Logs |
| I. | 6-week follow up assessment |
| J. | <b>End-of-treatment Assessment</b> |
| K. | 3-month, 6-month, 12-month follow up assessment |
| L. | Voucher Card |
| M. | <b>Drug Administration Subject Record</b> |
| N. | NRT Algorithm |
| 0. | <b>Stop Study Medication Profile</b> |
| <b>P.</b> | STOP Progress Note |
| Q. | STOP Prescription |
| R. | NRT Order Form-Pfizer |
| S. | NRT Internal Order Form |
| <b>T.</b> | Drug Shipment Record |
| U. | <b>Concomitant Medications Record</b> |
| V. | Signature and Delegation of Authority Log |
| W. | <b>Adverse Events Tracking Form</b> |
| <b>X.</b> | <b>Adverse Events Form</b> |
| <b>Y.</b> | Suspect Adverse Reaction Report |
| <b>Z.</b> | Pharmacy Card |
| AA. | Quality Control Form |
| BB. | Running Balance Inventory |

### **Attachments**

- 1. M.I.N.I.
- 2. LN.E.1 Venipuncture Procedure
- 3. STOP Brief Intervention Form
  Cigarette Withdrawal Scale
  Appointment Calendar
- 4. CAMH Delegation of Dispensing Policy
- 5. NRT Package Inserts
- 6. Cessation Resource List